CLINICAL TRIAL: NCT00079313
Title: A Pilot Study of the Safety and Efficacy of Imatinib in Reducing Monocytosis or Leukocytosis in Patients With Chronic Myelomonocytic Leukemia and Atypical Chronic Myelogenous Leukemia, Respectively
Brief Title: Imatinib (Gleevec(Registered Trademark)) to Treat Chronic Myelomonocytic Leukemia and Atypical Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Cynthia E. Dunbar, M.D./National Heart, Lung, and Blood Institute, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 040090; 04-H-0090; NCT00076297 (obsolete NCT alias)
Record Dates: First submitted 2004-03-08; First posted 2004-03-10 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-09-23

CONDITIONS: Chronic Myelomonocytic Leukemia; Chronic Myelogenous Leukemia
Keywords: CMML; CML; Gleevec; Glivec; STI-571; Tyrosine Kinase Inhibitor; Chronic Myelogenous Leukemia; Atypical Chronic Myelogenous Leukemia; Chronic Myelomoncytic Leukemia; Leukemia
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia | interventions — Imatinib Mesylate

INTERVENTIONS:
Drug: Imatinib

SUMMARY:
This study will evaluate the safety and effectiveness of imatinib (Gleevec(Registered Trademark)) in patients with chronic myelomonocytic leukemia (CMML) and atypical chronic myelogenous leukemia (CML). These conditions cause uncontrolled growth of malignant (cancerous) cells in the bone marrow that prevents the bone marrow from functioning normally in producing blood cells. The cancer cells also can spill over into the blood and invade other organs of the body. Imatinib has been approved by the Food and Drug Administration for treating chronic myelogenous leukemia, which has characteristics similar to atypical CML and to CMML, and data from other research suggests this drug may be able to produce a remission in forms of leukemia other than CML.

Patients over 18 years of age with atypical CML or CMML may be eligible for this study. Candidates are screened with a medical history and physical examination, blood tests, electrocardiogram, chest x-ray, and bone marrow aspiration and biopsy (removal of a small piece of bone marrow tissue through a needle inserted into the hip bone).

Participants take imatinib capsules once a day for 2 years. If at any time during the study the patient's blood counts begin to rise, disease symptoms develop, or the disease has progressed, the dose of imatinib is increased each week until the disease progression is stopped. Any patient whose disease does not response to treatment after 6 weeks of increased dosing and 30 days at the maximum daily dose of 800 mg is taken off the study and referred for different treatment.

Patients are seen by their referring physician every week for the first 4 weeks of the study, every other week for the next 8 weeks, and then monthly until the study is completed. At each visit, blood is drawn to monitor for drug side effects and response to therapy. In addition, patients come to the NIH Clinical Center every 3 months for a complete history and physical examination and for a bone marrow aspiration and biopsy every 6 months to assess the effect of treatment on bone marrow cells.

Patients who leave the study before 2 years are followed with laboratory monitoring for 6 months after stopping imatinib; those who remain on the drug for the full 2 years are monitored for 1 year after stopping the drug.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and effectiveness of imatinib for improving blood counts in patients with chronic myelomonocytic leukemia (CMML) and atypical chronic myelogenous leukemia (CML).

Although a number of agents have been used to treat these diseases, most patients do not respond to treatment. Imatinib has been shown in clinical trials to induce high rates of responses in patients with chronic phase CML. Imatinib has also been shown to be effective in inducing responses in a subset of patients with CMML and atypical CML and is also effective in a subset of patients with idiopathic hypereosinophilic syndrome (HES), another myeloproliferative disorder. Because patients with several different myeloproliferative diseases have been shown to experience dramatic responses to imatinib, we would like to determine what proportion of patients with atypical myeloproliferative diseases (CMML and atypical CML) will respond to this agent.

Prior to enrollment, a thorough clinical evaluation will be performed. A baseline bone marrow will be obtained to exclude acute leukemia or lymphoma and to assess the degree and nature of the myeloproliferation. In order to minimize bone marrow suppression, other myelosuppressive drugs will be tapered and discontinued during the first week of therapy with imatinib. Complete blood counts will be performed weekly for the first month and every other week thereafter. Clinical assessments will be performed every three months to assess for continued response.

ELIGIBILITY:
* INCLUSION CRITERIA:

All subjects must be greater than or equal to 18 years of age.

All subjects must meet the established diagnostic criteria for CMML or atypical CML.

The diagnostic criteria for CMML include:

* persistent peripheral blood monocytosis (greater than 1000/mm(3)),
* no Philadelphia chromosome or BCR/ABL fusion gene,
* fewer than 20% blasts in the blood and bone marrow, and
* dysplasia in one or more myeloid lineages. If dysplasia is absent the diagnosis of CMML can still be made if the other requirements are met and a cytogenetic abnormality is present in the marrow cells or if monocytosis has been persistent for at least 3 months and all other causes of monocytosis have been excluded.

OR

The diagnostic criteria for atypical CML include:

* peripheral blood leukocytosis comprised of increased mature and immature neutrophils,
* prominent dysgranulopoiesis,
* no Philadelphia chromosome or BCR/ABL fusion gene,
* neutrophil precursors greater than or equal to 10% of white blood cells,
* basophils less than 2% of white blood cells,
* monocytes less than 10% of white blood cells,
* hypercellular bone marrow with granulocytic proliferation and dysplasia, and fewer than 20% blasts in the blood and bone marrow.
* Serum creatinine less than 2mg/dl
* ECOG performance status less than 3
* Life expectancy greater than 12 weeks
* All subjects (men and women) must agree to practice abstinence or effective contraception during administration of imatinib.
* Patients must be able to comprehend the investigational nature of the research and be willing to sign an informed consent.

EXCLUSION CRITERIA:

Pregnancy or lactation.

HIV positivity or other known immunodeficiency.

Absolute neutrophil count less than 1000/mm(3) or platelet count less than 10,000/mm(3) or less than 50,000/m(3) with clinical evidence of bleeding.

Infection not adequately responding to appropriate therapy

History of non-hematologic malignancy treated with chemotherapy in past 5 years.

A moribund status or concurrent hepatic, renal, cardiac, metabolic disease of such severity that death within 12 weeks from initiation of therapy is likely.

Treatment with investigational agent (other than hematopoietic growth factors) within 4 weeks of study entry.

Psychiatric, affective, or other disorder that may compromise the ability to give informed consent or to cooperate in a research study.

Elevated transaminases (greater than 5 times the upper limit of normal) or elevated bilirubin (greater than 3 times the upper limit of normal).

Recent exposure to chickenpox or recent history of Herpes zoster (shingles) reactivation. Imatinib may put patients at increased risk of severe disease.

Left ventricular ejection fraction less than 45%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2004-01-14; Primary Completion 2006-12-30 (Actual); Study Completion 2010-10-25 (Actual)

PRIMARY OUTCOMES:
Peripheral blood absolute monocyte/leukocyte count measured at 2 months. | 2-months

SECONDARY OUTCOMES:
Resolution of bone marrow abnormalities, improvement in transfusion requirements, reduction or disappearance of cytogenetic abnormalities or fusion transcripts as detected by quantitative PCR/progression of clinical disease at 2 mths and every 3...

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Germing U, Gattermann N, Minning H, Heyll A, Aul C. Problems in the classification of CMML--dysplastic versus proliferative type. Leuk Res. 1998 Oct;22(10):871-8. doi: 10.1016/s0145-2126(97)00192-6. PMID 9766745
- [Background] Nosslinger T, Reisner R, Koller E, Gruner H, Tuchler H, Nowotny H, Pittermann E, Pfeilstocker M. Myelodysplastic syndromes, from French-American-British to World Health Organization: comparison of classifications on 431 unselected patients from a single institution. Blood. 2001 Nov 15;98(10):2935-41. doi: 10.1182/blood.v98.10.2935. PMID 11698274
- [Background] Fenaux P, Beuscart R, Lai JL, Jouet JP, Bauters F. Prognostic factors in adult chronic myelomonocytic leukemia: an analysis of 107 cases. J Clin Oncol. 1988 Sep;6(9):1417-24. doi: 10.1200/JCO.1988.6.9.1417. PMID 3166485